CLINICAL TRIAL: NCT03152279
Title: Assessment of Duodenal Epithelial Integrity in Celiac Disease With Mucosal Impedance
Status: Completed | Type: Observational
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Dhyanesh Patel, Principal Investigator, Vanderbilt University Medical Center
Other Study IDs: 161436
Record Dates: First submitted 2017-05-10; First posted 2017-05-15 (Actual); Last update posted 2021-05-06 (Actual); Status verified 2021-05

CONDITIONS: Celiac Disease
MeSH Terms: conditions — Celiac Disease | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Celiac Disease: Patients with suspected Celiac Disease who plan to undergo duodenal biopsy as part of routine clinical care
  Interventions: Diagnostic Test: Mucosal Impedance Catheter; Diagnostic Test: Blood sample
- Control: Patients scheduled for an upper endoscopy for indication other than evaluation of Celiac Disease or concern for CeD as part of routine clinical care
  Interventions: Diagnostic Test: Mucosal Impedance Catheter

INTERVENTIONS:
Diagnostic Test: Mucosal Impedance Catheter — During routine endoscopy, consented study participants will have a mucosal impedance catheter sensor positioned along the mucosal wall to measure resistance across the mucosa. The study procedure will add approximately 1-2 minutes of anesthesia time for each participant.
Diagnostic Test: Blood sample — At time of endoscopy, subjects with initial positive CeD serology will have a blood sample taken for any missing CeD serologies and intestinal fatty acid-binding protein (IFABP). This will be done at time of IV initiation as to avoid any additional venipuncture.
  Groups: Celiac Disease

SUMMARY:
Increased intestinal permeability can represent compromise of the epithelium's integrity and is thought to be the primary mechanism in patients who develop Celiac Disease (CeD) and non-celiac gluten sensitivity when gluten peptides cross the barrier and trigger an immune response. In this study, the investigators propose to use a novel, minimally invasive technology to detect mucosal damage (i.e. barrier dysfunction) in the duodenal epithelium. The primary aim of this study is to identify if there is a difference in duodenal mucosal impedance between CeD and control patients.

ELIGIBILITY:
Inclusion Criteria:

* scheduled for endoscopy as part of routine care with or without suspected Celiac Disease based upon at least 1 positive serologic marker of CeD
* consuming gluten at time of endoscopy

Exclusion Criteria:

* Already on a gluten free diet or unwilling to undergo a gluten challenge
* Undergoing upper endoscopy for an urgent indication such as unstable gastrointestinal bleed or food impaction
* Patients with inflammatory bowel disease
* Patients on blood thinners other than aspirin at time of endoscopy
* Patient unable to give informed consent
* Patient less than 18 years old

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Celiac disease patients will be identified in the Celiac Disease Clinic at Vanderbilt. Patients will be asked if they would like to participate in the study during their clinic visit and will undergo consent for the study at the time of procedure. Control subjects will be asked about participation at the time of routine endoscopy.
Sampling Method: Non-Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2018-11-07 (Actual); Study Completion 2018-11-14 (Actual)

PRIMARY OUTCOMES:
mucosal impedance values | Values will be obtained at conclusion of esophagogastroduodenoscopy (EGD), an expected average of 6 minutes
  Identify if there is a difference in duodenal mucosal impedance between CeD and control patients

SECONDARY OUTCOMES:
Marsh Score | 1 week
  Correlate measures of duodenal impedance with standardized pathology scores in CeD (Marsh Score)
IFABP | 1 week
  Identify whether there is a difference in IFABP in patients with normal and abnormal mucosal impedance

CONTACTS AND LOCATIONS:
Overall Officials: Dhyanesh Patel, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center Endoscopy Laboratory, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No